CLINICAL TRIAL: NCT04279197
Title: Efficacy and Safety of Fuzheng Huayu Tablets in Post-COVID-19 Patients With Pulmonary Inflammation and Fibrosis : A Multicenter Double-blind Randomized Controlled Trial
Brief Title: Treatment of Pulmonary Fibrosis Due to COVID-19 With Fuzheng Huayu
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Jingmen No.1 People's Hospital (Other); Wuhan No.1 Hospital (Other); Wuhan Third Hospital (Other); Huangshi Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Liu Chenghai, Institute Director, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fzhy-ncp-2
Record Dates: First submitted 2020-02-15; First posted 2020-02-21 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Fibrosis Due to COVID-19
MeSH Terms: interventions — fuzheng huayu; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FZHY Group (Experimental): usual treatment (respiratory function rehabilitation training + Vitamin C tablets)
  * Fuzheng Huayu tablets
  Interventions: Drug: Fuzheng Huayu Tablet; Drug: Vitamin C tablets; Other: respiratory function rehabilitation training
- Placebo Group (Placebo Comparator): usual treatment (respiratory function rehabilitation training + Vitamin C tablets)
  * placebo
  Interventions: Drug: Vitamin C tablets; Drug: Placebo; Other: respiratory function rehabilitation training

INTERVENTIONS:
Drug: Fuzheng Huayu Tablet — FZHY, administration: 0.4g/tablet, 1.6g/time, 3 times/day, oral; administered half an hour after the meal.
  Other Names: FZHY
  Arms: FZHY Group
Drug: Vitamin C tablets — Vitamin C tablets, administration: 0.2g/time, 3 times/ day, oral；
  Other Names: VC
Drug: Placebo — Placebo , administration: 0.4g/tablet, 1.6g/time, 3 times/day, oral; administered half an hour after the meal.
  Arms: Placebo Group
Other: respiratory function rehabilitation training — Health exercise, once a day

SUMMARY:
According to previous studies, viral pneumonia can develop into pulmonary fibrosis, which can affect patients'lung function and even life health.This study aims to observe the efficacy and safety of Fuzheng Huayu Tablets in the treatment of pulmonary fibrosis after COVID-19.

DETAILED DESCRIPTION:
The patients with COVID-19 could suffered from the pulmonary dysfunction and/or fibrosis the recovery period, but there are no certain drugs or treatment to cope with this situation. Our previous studies indicated that Fuzheng Huayu tablets (FZHY) could regress the lung fibrosis induced by bleomycin in animals, and improve the pulmonary function in the patients with chronic obstructive pulmonary disease. Now we design this trial to carry out the clinical study in order to evaluate the effects of Fuzheng Huayu tablets on pulmonary fibrosis and/or pulmonary function injury in the recovery period of COVID-19 and expect to improve the prognosis.

This is a randomized, double-blind, multicenter, placebo-controlled clinical trial.It enrolls 142 patients who had been diagnosed with COVID-19, but currently they are negative for viral testing and have developed pulmonary fibrosis or pulmonary dysfunction. They are randomly assigned into Placebo group and FZHY group. All patients are given usual treatment such as respiratory function rehabilitation training and vitamin C. The FZHY group is given Fuzheng Huayu tablets, and the control group is given placebo. Each patient will be observed for 24 weeks and followed up for 8 weeks. The primary outcomes for the trial are the improvement proportion of pulmonary fibrosis judged by HRCT score and the improvement of lung function(FVC,FEV1,FVC/FEV1). Secondary outcomes include six-minute walk distance, improvement proportion of pulmonary inflammation, improvement proportion of clinical symptoms , quality of Life-BREF (QOL-BREF) Score, patient health questionnaire-9 (PHQ-9) Score, general anxiety disorder-7 (GAD-7) score. The safety also be observed.

ELIGIBILITY:
Inclusion criteria (I) Discharged patients fulfilling the diagnostic criteria of COVID-19 (China Diagnosis and Treatment Protocol for COVID-19 (Trial Version 7); (II) COVID-19 RNA in respiratory specimens or blood specimens of patients is negative (>2 times), assayed by real-time fluorescent polymerase chain reaction test (RT-PCR); (III) Pulmonary CT scans within 7 days showed that there were still unabsorbed inflammation or pulmonary fibrosis in the lungs; (IV) Age 18-70.

Exclusion criteria

* Patients who have undergone lung surgery that affects pulmonary function, such as pulmonary transplantation, pulmonary resection, pulmonary volume reduction, etc;
* Relying on mechanical ventilation to maintain pulmonary function, such as ventilators;
* Combined with chronic pulmonary diseases affecting pulmonary function, such as chronic obstructive pulmonary disease, other known causes of interstitial pulmonary disease;
* Patients with diseases affecting cardiac function, such as pulmonary circulation hypertension, heart failure, peripheral vascular disease, fibromyalgia, and pacemaker installation;
* Patients with severe underlying diseases affecting survival, including uncontroled cardiac, renal, digestive, hematological, neuropsychiatric, immune, metabolic diseases, malignant diseases and severe malnutrition;
* Resting heart rate >120 times/min;
* Systolic blood pressure > 180 mmHg, diastolic blood pressure > 100 mmHg;
* Unstable angina pectoris or myocardial infarction occurring within the last month;
* Severe obesity (BMI > 30 kg/m2);
* Allergic constitution, allergic to the drug components involved in the treatment program;
* Pregnant or breastfeeding women;
* Patients with disabilities who are unable to complete the efficacy evaluation questionnaires;
* Difficult collaborators with poor mental health status, suffering from mental illness, patients without self-control, unable to express clearly;
* Those who are participating in other clinical trials;
* According to the investigator's judgment, patients whose enrollment complications or poor compliance will affect the efficacy and safety evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
The improvement proportion of pulmonary fibrosis | Week 24
  Evaluation of pulmonary fibrosis Improvement. pulmonary fibrosis judged by HRCT score.HRCT images are divided into four grades according to the score, and a reduction of one grade is an improvement.
The improvement of lung function | Week 24
  FVC, FEV1, FVC/FEV1

SECONDARY OUTCOMES:
The improvement proportion of pulmonary inflammation | Week 24
  Evaluation of pulmonary inflammation Improvement
The improvement proportion of clinical symptom | Week 24
  Discomfort symptoms include dyspnea, cough, exhausted, fatigue, insomnia, sweating, poor appetite, diarrhea, etc., which are common manifestations of patients with COVID-19
Quality of Life-BREF (QOL-BREF) | Week 24
  This scale can reflect the quality of life of patients to some extent.
Patient Health Questionnaire-9(PHQ-9) | Week 24
  This scale can reflect the quality of life of patients to some extent.
Generalized anxiety disorder-7(GAD-7) | Week 24
  This scale can reflect the quality of life of patients to some extent.
The 6-minute walk distance | Week 24
  Evaluation of Lung Function Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Chenghai Liu, Study Director — Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shuguang Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jing F, Wang W, Ke J, Huang T, Jiang B, Qiu Q, Huang J, Zhan S, Zhang W, Wu H, Su W, Feng J, Peng Y, Zhao Z, Xing F, Liu C. Fuzheng Huayu tablets for treating pulmonary fibrosis in post-COVID-19 patients: a multicenter, randomized, double-blind, placebo-controlled trial. Front Pharmacol. 2025 Mar 11;16:1508276. doi: 10.3389/fphar.2025.1508276. eCollection 2025. PMID 40135237